CLINICAL TRIAL: NCT02488590
Title: Systematic Approach for the Diagnosis and Treatment of Obstructive Lung Diseases
Acronym: ACOS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Wim Janssens, Prof. Dr. Wim Janssens, KU Leuven
Other Study IDs: S57767
Record Dates: First submitted 2015-06-29; First posted 2015-07-02 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Chronic Obstructive Pulmonary Disease; Asthma; Overlap Syndrome
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma | interventions — laminin A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- CHRONIC OBSTRUCTIVE PULMONARY DISEASE: Patients with an obstructive spirometry and characteristics of chronic obstructive pulmonary disease
  Clinical intervention:
  Long acting B agonist (LABA) + Long acting muscarinic receptor antagonist (LAMA) inhaled therapy
  Interventions: Drug: LABA + LAMA
- ASTHMA: patients with asthma and a normal spirometry
  Clinical intervention: Inhaled corticosteroids (ICS)
  Interventions: Drug: ICS
- ASTHMA COPD OVERLAP SYNDROME: patients with an obstructive spirometry and characteristics of both COPD and Asthma
  Clinical Intervention: LABA + LAMA + ICS
  Interventions: Drug: LABA + LAMA + ICS
- OBSTRUCTIVE ASTHMA: patients with an obstructive spirometry and characteristics of asthma
  Clinical Intervention: LABA + ICS inhaled therapy
  Interventions: Drug: LABA + ICS
- OTHER: patients with another diagnosis or healthy persons
  clinical Intervention: undefined - according to diagnosis
  Interventions: Drug: other

INTERVENTIONS:
Drug: LABA + LAMA — An open label inhaled therapy is initiated once the diagnosis has been set based on clinical and testing criteria (algorithm). The treatment may be changed in function of the clinical evolution, which is left at the discretion of the general practitionar. Changes in treatment and treatment doses are registered during 1 year follow-up.
  Other Names: dual bronchodilation
  Groups: CHRONIC OBSTRUCTIVE PULMONARY DISEASE
Drug: ICS — An open label inhaled therapy is initiated once the diagnosis has been set based on clinical and testing criteria (algorithm). The treatment may be changed in function of the clinical evolution, which is left at the discretion of the general practitionar. Changes in treatment and treatment doses are registered during 1 year follow-up.
  Other Names: inhaled cortiscosteroids
  Groups: ASTHMA
Drug: LABA + LAMA + ICS — An open label inhaled therapy is initiated once the diagnosis has been set based on clinical and testing criteria (algorithm). The treatment may be changed in function of the clinical evolution, which is left at the discretion of the general practitionar. Changes in treatment and treatment doses are registered during 1 year follow-up.
  Other Names: triple therapy
  Groups: ASTHMA COPD OVERLAP SYNDROME
Drug: LABA + ICS — An open label inhaled therapy is initiated once the diagnosis has been set based on clinical and testing criteria (algorithm). The treatment may be changed in function of the clinical evolution, which is left at the discretion of the general practitionar. Changes in treatment and treatment doses are registered during 1 year follow-up.
  Other Names: bronchodilator inhaled corticosteroid fixed combinations
  Groups: OBSTRUCTIVE ASTHMA
Drug: other — An open label therapy or no therapy is initiated once the diagnosis has been set based on clinical and testing criteria (algorithm). The treatment may be changed in function of the clinical evolution, which is left at the discretion of the general practitionar. Changes in treatment and treatment doses are registered during 1 year follow-up.
  Other Names: no inhalation therapy
  Groups: OTHER

SUMMARY:
The differential diagnosis of asthma and COPD is sometimes difficult. Recently, an overlap syndrome has been defined based on the concurrence of asthma and COPD characteristics. These characteristics are based on expert opinions and have never been investigated nor validated prospectively.

The investigators assume that the management strategy, the symptom burden and disease progression will differ between asthma, COPD and ACOS. Therefore, the study wants to establish baseline criteria for an appropriate disease definition and evaluate the potential impact on treatment and symptom control.

DETAILED DESCRIPTION:
This study aims to test a diagnostic algorithm for obstructive airways diseases that may be used in daily practice to obtain a correct differential diagnosis and, hence, initiate an adequate therapy according to the current guidelines. The proposed algorithm will be used to categorize patients in 4 different diagnoses with specific treatment choices: asthma, obstructive asthma, overlap asthma with COPD, and COPD. The study will evaluate which tests and criteria contribute most to the diagnostic work-up and final diagnosis.

Test battery for diagnosis

* spirometry with bronchodilator reversibility testing
* bodyplethysmography: spirometry, volumes, resistance, diffusing capacity
* exhaled NO
* blood sample
* CT scan of thorax (only when obstructive spirometry)
* histamine challenge (only when spirometry is not obstructive)
* induced sputum (not for protocol interpretation)

Definition of endpoints

1. Physician based diagnosis:

   diagnosis based on clinical exam and spirometry
2. Algorithm based diagnosis:

   diagnosis based on clinical exam and test battery
3. Final standard diagnosis diagnosis based on clinical exam, test battery and clinical evolution of 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with respiratory symptoms suggestive of chronic airway disease

Exclusion Criteria:

* Subjects with an immediate need for hospitalization or a treatment of systemic glucocorticoid or long-term antibiotics
* Subjects with pregnancy
* Subjects with clinically significant cardiovascular disease that warrants intervention
* Subject with concomitant pulmonary diseases (pulmonary embolism, interstitial lung disease etc..).

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients of Caucasian descent, ageing 30-80 years and presenting for the first time at the outpatient pulmonary clinic of the University Hospitals Leuven with respiratory symptoms
Sampling Method: Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2015-07; Primary Completion 2020-04 (Actual); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Accuracy of the proposed diagnostic algorithm | after work-up at inclusion (at baseline)
  % changes of algorithm diagnosis compared to physician based diagnosis (based on spirometry only)
Accuracy of the proposed diagnostic algorithm (at one year follow-up) | at one year
  % changes of algorithm diagnosis compared to final diagnosis (based on all tests with clinical evolution for 1 year))

SECONDARY OUTCOMES:
Difference in ACT/CAT-scores | 3 months
  Difference of ACT/CAT-score between arms at 3 months
Difference in ACT/CAT-scores | 1 year
  Difference of ACT/CAT-scores between arms at 1 year
Difference in Delta ACT/CAT scores (0 - 3 months) | 3 months
  Difference of delta ACT/CAT-scores (0 - 3 months) between arms
Difference in Delta ACT/CAT scores (0 - 1 year) | 1 year
  Difference of delta ACT/CAT-scores (0 - 1 year) between arms
specificity and sensitivity of individual criteria for final diagnosis | 1 year
  ROC curve analysis for individual criteria in predicting final diagnosis
independency of criteria for final diagnosis | 1 year
  Logistic regression analysis for criteria in predicting final diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Wim Janssens, MD, Principal Investigator — KU Leuven
Locations (1):
- UZ Gasthuisberg, Leuven, Flanders, Belgium